CLINICAL TRIAL: NCT02695758
Title: Local Intraoperative Analgesic Injection Versus Single Injection Interscalene Nerve Block in Patients Undergoing Shoulder Arthroplasty (TSA): A Randomized Trial
Brief Title: Local Intraoperative Analgesic Injection Versus Single Injection Interscalene Nerve Block in Patients Undergoing TSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016Nam2
Record Dates: First submitted 2016-02-22; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Osteoarthritis: Shoulder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- interscalene brachial plexus block (Active Comparator): Direct interscalene nerve block injection via brachial plexus
  Interventions: Procedure: Interscalene brachial plexus block
- Bupivacaine extended-release liposome injection (Active Comparator): Infiltration of local anesthetic/analgesic, Bupivacaine extended-release liposome injection (Exparel) + Diluted in 40cc of Saline into the capsule, subscapularis, deltoid, pectoralis major and subcutaneous tissues.
  Interventions: Procedure: bupivacaine extended-release liposome injection

INTERVENTIONS:
Procedure: Interscalene brachial plexus block
  Arms: interscalene brachial plexus block
Procedure: bupivacaine extended-release liposome injection
  Arms: Bupivacaine extended-release liposome injection

SUMMARY:
A non-blinded randomized controlled trial, in which participants undergoing primary reverse or total shoulder arthroplasty are randomly assigned to one of two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. All individuals undergoing primary reverse and total shoulder arthroplasty by the shoulder service at Methodist Hospital or Rothman Specialty Hospital.

Exclusion Criteria:

1. Psychiatric illness as defined by co-morbid diagnosis of bipolar disorder or schizophrenia
2. Revision arthroplasty, arthroplasty for fracture
3. Unable/unwilling to consent for enrollment
4. Unable to complete postoperative pain survey
5. Known adverse drug reaction or allergy to the medications used
6. Chronic pain syndromes (including reflex sympathetic dystrophy, fibromyalgia, chronic diffuse musculoskeletal pain)
7. Patients taking long acting narcotic pain medications (including extended release narcotic pain medications and methadone).
8. Patients under the age of 18 years
9. Patients with history of hepatic disease
10. Pregnant women or women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Morphine and Morphine Equivalent consumption | 24 hours following surgery